CLINICAL TRIAL: NCT05289921
Title: Multi Center, Phase III Clinical Trial to Evaluate the Safety and Efficacy of LIZTOX Inj in the Treatment of Post Stroke Upper Limb Spasticity
Brief Title: To Evaluate HU-014 in the Treatment of Post Stroke Upper Limb
Acronym: HU-014
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-014_P3_ULS
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Post Stroke Upper Limb Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HU-014 Inj (Experimental): HU-014 Inj was given an injection to 5 Upper limb muscle(Total 360U/, IM)
  Interventions: Biological: HU-014 Inj
- Clostridium botulinum type A (Active Comparator): Clostridium botulinum type A Inj was given an injection to 5 Upper limb muscle(Total 360U/, IM)
  Interventions: Biological: HU-014 Inj

INTERVENTIONS:
Biological: HU-014 Inj — HU-014 Inj was given an injection to 5 Upper limb muscle

SUMMARY:
Investigational Product: LIZTOX inj 100unit(HU-014) Title : Multi Center, Phase III Clinical Trial to Evaluate the efficacy and Safety of LIZTOX Inj in the Treatment of Post Stroke Upper Limb Spasticity Sites and investigators : Asan Medical Center(Seoul), Min-ho Chun, M.D, Ph.D Objective : To evaluate the efficacy and safety of LIZTOX inj in the treatment of Post Stroke Upper Limb Spasticity

ELIGIBILITY:
Inclusion Criteria:

* A subject who is diagnosed with Stroke at least six weeks prior to Screening.
* A subject who has Modified ashworth scale(MAS) score which Wrist Flexor is ≥ 2 and Flexor or Finger Flexor is ≥ 1.
* A subject with a Disability assessment scale(DAS)of at least ≥ 2 in one of the categories of hand hygiene, clothing, upper extremity, or pain for evaluation.

Exclusion Criteria:

* A subject who has medical history following. (Allergy, Chemodenervation(within 6 months), Tendon lengthening(within 6 months), Intrathecal baclofen.Aspiration pneumonia, etc.)
* A subject who has history of any diseases following. (neuromuscular junction disorder, NMJ, myasthemia gravis, MG, Lambert-Eaton myasthenic syndrome, amyotrophic lateral sclerosis, ALS, Skin disease, Dysphagia, etc.)
* From screening, Subject who get a plastic Surgery including fascioplasty, Prosthesis implantation within 6 Weeks
* Subject who takes a medication including skeletal muscle relaxants, Aminoglycoside, lincomycin, anticholinergic drug, benzodiazepine, benzamide etc.
* A subject who tend to bleed or are taking anti-coagulant drugs.
* A sugject who is undergoing rehabilitation(physical therapy, occupational therapy, exercise therapy) or Splinting in the area where medication for clinical trials is scheduled to be administered.
* A sugject who has muscle atrophy, fixed joint/muscle contracture in the area where medication for clinical trials is scheduled to be administered.
* Any condition that, in the view of the investigator, would interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
MAS score improvement at Wrist Flexor | 4 weeks
  The rate of change in muscle tension measured by MAS

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea